CLINICAL TRIAL: NCT06645561
Title: Radiological Dating of Child Fractures Before One Year
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 23-HPNCL-02
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-02

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants under one year
  Interventions: Procedure: X-ray

INTERVENTIONS:
Procedure: X-ray — defined radiographic semiological criteria to determine an analytical methodology to facilitate the dating of long bone fractures of infants under one year of age

SUMMARY:
The aim of this study was to use, in a precise manner, defined radiographic semiological criteria to determine an analytical methodology to facilitate the dating of long bone fractures of infants under one year of age. A total of 99 radiographs of infants under one year of age with long bone fractures of known date were studied. Four dating groups were established on the basis of data in the literature, with the aim of developing predictive models based on well-defined semiological criteria, in order to construct a simplified dating decision tree.

ELIGIBILITY:
Inclusion Criteria:

* had X-rays taken at the University Paediatric Hospital for the diagnosis and/or follow-up of a fracture of the long bones of the limbs (tibia, femur, fibula, radius, humerus and/or ulna)

Exclusion Criteria:

* child maltreatment,
* chronic illnesses

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 99 radiographs of infants under one year of age with long bone fractures of known date were studied.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Dating fracture | between 2011 and 2023
  in days

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Lenval, Nice, France